CLINICAL TRIAL: NCT01826409
Title: Hypoglycemic Effects of Fermented Red Ginseng in Subject With Impaired Fasting Glucose or Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WKP-FG7070-001
Record Dates: First submitted 2013-04-04; First posted 2013-04-08 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Impaired Glucose or Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fermented red ginseng (Experimental)
  Interventions: Dietary Supplement: Fermented Red Ginseng
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented Red Ginseng — Fermented red ginseng 2.7g/day for 4 weeks
  Arms: Fermented red ginseng
Dietary Supplement: Placebo — Placebo 2.7g/day for 4 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of fermented red ginseng (FRG) on glycemic status in subjects with impaired fasting glucose (IFG) or type 2 diabetes.

DETAILED DESCRIPTION:
This study was a 4 weeks, randomized, double-blind, placebo-controlled trial. Forty-two subjects with IFG or type 2 diabetes were randomly allocated to 2 groups to consume placebo or FRG three times per day for 4 weeks. Fasting and postprandial glucose profiles during meal tolerance test were assessed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years with fasting glucose 100~140 mg/dL at least two of the following

Exclusion Criteria:

* Lipid metabolic disorder
* Acute or chronic inflammatory disease
* Taking medication of corticosteroid within 4 weeks of the study
* Cardiovascular disease (arrhythmia, heart failure, myocardial infarction or patient with pacemaker)
* Allergic or hypersensitive to any of the ingredients in the test products
* Participation in other clinical trials within 2 months
* Abnormal hepatic liver function or renal disease (acute/chronic renal failure or nephrotic syndrome)
* Taking medication of lipid phosphates within 3 months of the study etc,

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Glucose profiles during meal tolerance test | 4 weeks
  Fasting and postprandial glucose profiles during meal tolerance test were assessed before(baseline) and after the intervention

SECONDARY OUTCOMES:
Change in lipid profiles | 4 weeks
  Change in lipid profiles were assessed before(baseline) and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tae Sun Park, MD., PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clincial Trial Center for Functional Foods, Jeonju, Jeollabok-do, South Korea

REFERENCES:
- [Derived] Oh MR, Park SH, Kim SY, Back HI, Kim MG, Jeon JY, Ha KC, Na WT, Cha YS, Park BH, Park TS, Chae SW. Postprandial glucose-lowering effects of fermented red ginseng in subjects with impaired fasting glucose or type 2 diabetes: a randomized, double-blind, placebo-controlled clinical trial. BMC Complement Altern Med. 2014 Jul 11;14:237. doi: 10.1186/1472-6882-14-237. PMID 25015735